CLINICAL TRIAL: NCT07081893
Title: Development of the PEC-REHAB Instrument: Enhancing and Measuring Person-Centeredness in Rehabilitation Services, a Qualitative Study
Brief Title: How do Patients, Relatives and Healthcare Professionals View Person-centered Rehabilitation.
Acronym: PECRehab
Status: Not yet recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Liselot Thijs, dr, Hasselt University
Other Study IDs: Patient centered rehab
Record Dates: First submitted 2025-07-07; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Patient Centered Care
Keywords: Patient centered care; Healthcare professionals; Perspective; Relatives; Patients; Rehabilitation; Students
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthcare professionals: This cohort includes healthcare professionals who are actively working within a rehabilitation center or rehabilitation department. Eligible participants are aged 18 years or older and have provided written informed consent. No active interventions are performed in this study. Participants are invited to take part in a focus group or an in-depth interview to share their experiences and perspectives related to person-centered care in rehabilitation.
  Interventions: Other: Conventional care with semi-structured interviews and focus groups
- Patients and relatives involved in a rehabilitation process: This cohort includes individuals who are currently admitted to a rehabilitation center or rehabilitation department, as well as relatives or close contacts of such patients. Eligible participants are aged 18 years or older and have provided written informed consent. No active interventions are performed in this study. Participants are invited to take part in an in-depth interview to share their experiences and perspectives related to person-centered care in rehabilitation.
  Interventions: Other: In-depth interviews with patients and relatives
- Students doing an internship in a rehabilitation department or centre: This cohort includes students linked with an education within a healthcare profession. The students did an actively internship within a rehabilitation center or rehabilitation department. Eligible participants are aged 18 years or older and have provided written informed consent. No active interventions are performed in this study. Participants are invited to take part in a focus group or an in-depth interview to share their experiences and perspectives related to person-centered care in rehabilitation.
  Interventions: Other: Conventional care with additional focusgroups
- Board members, staff members and representatives: This cohort includes board members, staff members and representatives who are actively working within a rehabilitation center or rehabilitation department. Eligible participants are aged 18 years or older and have provided written informed consent. No active interventions are performed in this study. Participants are invited to take part in a focus group or an in-depth interview to share their experiences and perspectives related to person-centered care in rehabilitation.
  Interventions: Other: Semi-structured interviews and focus groups

INTERVENTIONS:
Other: Conventional care with semi-structured interviews and focus groups — In semi-structured individual interviews, employees of healthcare organisations are asked about their experiences, opinions and knowledge on person-centredness. This makes it possible to gather in-depth insights. This approach will mainly be used when surveying e.g. board members, managers, representatives of patient organisations. In addition, focus groups (6 to 8 people) will be organised. This is especially valuable when surveying doctors, paramedics and nurses. Focus groups make it possible to survey several respondents at the same time, encourage spontaneous conversations and share experiences. The interaction between participants can also ensure that additional perspectives and insights are covered.
  Groups: Healthcare professionals
Other: In-depth interviews with patients and relatives — The objective is to thoroughly understand what PEC means in rehabilitation. Although PEC can be understood as 'being responsive to the unique wishes and needs of the individual person', there still is a lack of consensus about its exact conceptualization in the rehabilitation context (Yun and Choi 2019). Prior work often only considers PEC in terms of shared decision making and goal setting, while the holistic perspective on the patient as a whole person is largely neglected (Yun and Choi 2019). This qualitative phase thus focuses on understanding PEC, its dimensions and the unique wishes and needs of patients in rehabilitation services. In addition, we gather insights regarding the potential enhancement of PEC in rehabilitation. The interviews are based on the Trajectory Touchpoint Technique (TTT; Sudbury-Riley et al. 2020a; 2020b) which allows us to uncover the unique experiences of respondents (i.e., patients, relatives, informal caregivers). The TTT is especially suited fo
  Groups: Patients and relatives involved in a rehabilitation process
Other: Semi-structured interviews and focus groups — In semi-structured individual interviews, employees of healthcare organisations are asked about their experiences, opinions and knowledge on person-centredness. This makes it possible to gather in-depth insights. This approach will mainly be used when surveying e.g. board members, managers, representatives of patient organisations. In addition, focus groups (6 to 8 people) will be organised. This is especially valuable when surveying doctors, paramedics and nurses. Focus groups make it possible to survey several respondents at the same time, encourage spontaneous conversations and share experiences. The interaction between participants can also ensure that additional perspectives and insights are covered.
  Groups: Board members, staff members and representatives
Other: Conventional care with additional focusgroups — In semi-structured individual interviews, students of healthcare organisations are asked about their experiences, opinions and knowledge on person-centredness. The focus groups will be supported by the Lego® Serious Play (LSP) will be used to collect in-depth insights from students. This design allows flexibility in questioning, while still following a consistent structure to explore common themes across focus groups. The use of Lego encourages participants to think in new ways.
  Groups: Students doing an internship in a rehabilitation department or centre

SUMMARY:
This research project aims to integrate insights from marketing and rehabilitation sciences to investigate Person Centered in rehabilitation.

The research objectives are

1. to better understand what Person Centered Rehabilitation means in rehabilitation,
2. to understand how Person Centered Rehabilitation can be enhanced
3. to develop an instrument that can be used as a quality indicator to evaluate and monitor Person Centered Rehabilitation in rehabilitation
4. to understand the impact of Person Centered Rehabilitation on key outcomes in rehabilitation.

To recruit respondents, we will work together with different rehabilitation centers and hospitals with a rehabilitation department.

The interviews will be based on the Trajectory Touchpoint Technique. The interviews will be transcribed and uploaded in NVivo 14. To code the data, we will use the Gioia method which offers a systematic approach to bring qualitative rigor in qualitative research and contains of four steps.

1. We will code the data based on first-order terms.
2. we will systematically examine these first-order terms to organize them into second-order theory-centric themes.
3. we will investigate whether it is possible to categorize the second-order themes into aggregate dimensions which serve to summarize the key components of the emerging theory
4. when we have the full set of first-order terms, second-order themes and aggregate dimensions, we will have all ingredients for building a data structure. The data structure provides a graphical presentation of how we progressed from raw data to themes and dimensions.

DETAILED DESCRIPTION:
Person-centeredness (PEC) has emerged as a key concept in modern healthcare, marking a shift away from disease-centered models toward approaches that acknowledge and respond to the unique needs, wishes, and contexts of each individual. Within rehabilitation services, this holistic orientation is especially pertinent, given the complex interplay between physical, emotional, psychological, and social factors influencing recovery and reintegration into daily life.

Despite growing recognition of its importance, PEC remains under-defined and insufficiently operationalized in rehabilitation settings. Current efforts to assess PEC tend to focus on outcomes such as patient satisfaction or functional status, rather than directly measuring the degree to which care is aligned with individual needs and preferences. A valid and reliable measurement instrument to evaluate PEC from the patient's perspective is currently lacking.

This study addresses that gap by developing the PEC-REHAB instrument. It aims to conceptualize PEC in rehabilitation, identify its key dimensions, explore ways to enhance PEC, and ultimately validate a tool to serve as a quality indicator. This protocol describes the second step of the qualitative phase of the study, which consists of in-depth interviews with patients and their informal caregivers.

The qualitative research follows a two-step structure:

1. Interviews and focus groups with rehabilitation care professionals.
2. In-depth interviews with patients and their relatives.

Data collection in this second step uses the Trajectory Touchpoint Technique (TTT)-a person-centered qualitative methodology that helps respondents articulate their lived experiences through visual prompts representing key stages of the rehabilitation journey. These stages include:

* First symptoms
* Pre-arrival planning
* Admission
* Stay in the rehabilitation center or department
* Discharge and aftercare

Each stage is represented by a laminated picture card showing various potential touchpoints. Respondents are encouraged to use these cards flexibly to narrate their experiences, ensuring a comprehensive yet personalized account of their rehabilitation journey. The TTT approach fosters inclusivity, reduces interviewer bias, and enhances respondent engagement.

The interviews also include semi-structured questions focused on:

* Respondents' understanding and experience of person-centeredness
* Perceived gaps and areas for improvement in PEC delivery
* The perceived importance and impact of PEC on well-being

All interviews will be audio-recorded with consent and transcribed verbatim. Data analysis will follow the Gioia methodology, a rigorous approach to qualitative coding that progresses through:

1. First-order coding based on respondents' own words
2. Development of second-order theory-based themes
3. Aggregation into overarching dimensions
4. Creation of a structured data model to inform theory development

Insights derived from this qualitative phase will directly inform the design and content of the PEC-REHAB instrument. The tool will be validated in a subsequent quantitative phase and used to assess whether rehabilitation services align with person-centered care principles from the patient's perspective.

Ultimately, this research aims to support the implementation of PEC in rehabilitation, provide actionable quality indicators, and contribute to improved outcomes by ensuring that rehabilitation services respond to the individuality of each patient.

ELIGIBILITY:
Patients and relatives

Inclusion Criteria:

* (1) are or were admitted to a rehabilitation centre or is related/ acquainted with someone admitted to a rehabilitation centre
* (2) are older than 18 years
* (3) speak the Dutch language
* (4) suffer from a non-congenital brain injury, neurological or locomotor condition can participate in this study.

Exclusion Criteria:

(1) did not sign informed consent

Healthcare professionals and board members, staff members and representatives

Inclusion Criteria:

1. are employed at a rehabilitation centre
2. are older than 18 years
3. speak the Dutch language

Exclusion Criteria:

(1) did not sign informed consent

Healthcare students

Inclusion Criteria:

1. did internships in a rehabilitation centre
2. are older than 18 years
3. speak the Dutch language

Exclusion Criteria:

(1) did not sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rehabilitation centers in Flanders
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Definition of Person-centered rehabilitation. | From start study to end of study, an average of 1 year
  Open-ended responses to the research questions; What is PEC in rehabilitation?
  No fixed measurement scale is used. Responses are analyzed using the Gioia method, resulting in a data structure based on first-order terms, second-order themes, and aggregate dimensions.

SECONDARY OUTCOMES:
What are the dimensions of person-centered rehabilitation | From start study to end of study, an average of 1 year
  Open-ended responses to the research questions; Which PEC dimensions (i.e., unique wishes and needs) can we discern in rehabilitation? No fixed measurement scale is used. Responses are analyzed using the Gioia method, resulting in a data structure based on first-order terms, second-order themes, and aggregate dimensions.
How can person-centered rehabilitation be enhanced? | From start study to end of study, an average of 1 year
  Open-ended responses to the research questions; How can PEC be enhanced? No fixed measurement scale is used. Responses are analyzed using the Gioia method, resulting in a data structure based on first-order terms, second-order themes, and aggregate dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Lamers, PhD, Principal Investigator — UHasselt

IPD SHARING:
Plan to Share IPD: No
This research is mainly organised in focus groups and interviews. Sharing individual data is therefore very difficult.